CLINICAL TRIAL: NCT06624267
Title: Small Vessel Disease of the Brain and Heart: a Perfusion PET Study of Training Effects
Brief Title: Test of Reproducibility of [15O]H20-PET Assessment of Brain Perfusion
Acronym: SVAT
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Danish Cardiovascular Academy (Unknown); Bispebjerg Hospital (Other); The Dagmar Marshall Foundation (Other); Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Thomas Ehlig Hjermind Justesen, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: H-24052476; PhD2024013-HF (Other Grant/Funding Number: Danish Cardiovascular Academy)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Microvascular Disease; Microvascular Complications; Diabetes Mellitus Type 2; Cerebral Hypoperfusion; Dementia
Keywords: microvascular disease; microvascular complications of the heart; microvascular complications of the brain; microvascular disease patophysiology; diabetes type 2; dementia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 24 healthy participants over 60 years: Baseline measurements of: -[15O]H2O PET of the brain
  Interventions: Diagnostic Test: PET

INTERVENTIONS:
Diagnostic Test: PET — PET imaging will be performed with a Discovery 710 PET/CT scanner (GE Healthcare, Milwaukee, WI, USA). Two 5-minute PET recordings will be performed of each subject within a single scanning session of 70 min. One 5-minute scan is conducted of the brain in rest. [15O]H2O, is produced on-site (GENtrace, GE, Uppsala, Sweden), and 600 MBq [15O]H2O is intravenously injected by an automatic Hidex Radiowater Generator (Hidex, Turku, Finland). To induce brain vasodilation, 1 g of acetazolamide is infused over 5 min and 15 min later the brain is scanned. Cerebral perfusion is calculated using PMOD software (PMOD Technologies, Switzerland).

SUMMARY:
In the aging population, ischemic heart disease, stroke and dementia are increasingly prevalent. Diagnosis and treatment of the former two i.e., large-vessel coronary heart disease and endovascular thrombectomy of the brain in relation to stroke have improved significantly. Yet, the majority of elderly patients with ischemic heart disease do not have large-vessel heart disease and it seems that small vessel disease (SVD) may explain a large fraction of these cases as well as the cardiovascular morbidity in the elderly. Hence, the current development in diagnostics and treatments of ischemic heart disease does not address the most common subtype of ischemic disease seen in elderly patients.

It has been suggested that SVD is part of a multisystem disorder and several systematic reviews have addressed the hypothesis of a potential link between small vessel disease of the heart, brain, and kidneys. Cerebral SVD is prevalent in the aging population causing cognitive impairment, dementia, and an increased risk of stroke, and cerebral hypoperfusion is an acknowledged cause of vascular dementia and a possible cause of Alzheimer's disease. Further, cognitive impairment within multiple cognitive domains is highly prevalent in heart failure and is associated to an increased risk of dementia. The link between heart failure and dementia may be due to multisystem SVD, although a direct link between the two is possible.

Among other known risk factors such as age, hypertension, and female sex, diabetes is a major cause of SVD and is linked to coronary heart disease as well as cognitive impairment. The diagnosis of cerebral SVD relies on MRI detecting infarctions, haemorrhages, microbleeds and ischemic white matter changes, i.e. Fazekas score. In contrast, perfusion PET is used to image myocardial perfusion in patients with coronary SVD; and coronary SVD is recognized as a part of the pathophysiology in angina, coronary artery disease, and heart failure. Perfusion PET before and after adenosine-induced vasodilation allows for measuring, the myocardial flow reserve (MFR), i.e. perfusion capacity, which in the absence of regional perfusion defects, is a measure of coronary SVD. Prof. Eva Prescott have recently shown that reduced MFR obtained by 82Rb PET is a strong predictor of future microvascular events and all-cause mortality.

Exercise is well known to improve cognitive health but professor Carl-Johan Boraxbekk has shown that the effect on cognitive performance may be dependent on the initial cerebrovascular status, as patients with moderate to severe white matter changes did not improve after a 6 months physical activation intervention in contrast to patients with mild changes. Yet, it is possible to improve brain function in diabetic patients through either dietary or exercise interventions.

Systemic SVD is measured as cerebral SVD (reduced brain perfusion during acetazolamide-induced vasodilation) and coronary SVD (reduced heart perfusion during adenosine-induced vasodilation). The researchers anticipate that patients with type 2 dabetes have reduced perfusion capacity of the brain and heart correlating to reduced cognition and cardiorespiratory fitness (VO2-max).

DETAILED DESCRIPTION:
The researchers wish to test how large the variance of their measurements of blood perfusion to the brain is in healthy participants when performing 2 identical examinations within 7 days of each other.

To adress this aim the researchers have defined the following assumption that they will refute or confirm through their study:

- PET-perfusion measurements at their department have a high reproducibility.

8 healthy participants over 60 years will undergo a [15O]H2O-PET scan in order to assess the blood perfusion capacity of the brain.

Within 7 days, the 8 healthy participants will undergo an additional [15O]H2O-PET scan assessing the blood perfusion capacity of the brain.

Afterwards the researchers will quantify the variance in their [15O]H2O-PET scan in the same individuals within a 7-day time window.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* No diagnosis of T2D according to WHO's criteria.
* Speaks and understands Danish (required for reliable cognitive testing)
* Able to provide informed and written consent

Exclusion Criteria:

* Moderate to high intensity training >2 times/week.
* Previous AMI, atrial fibrillation, significant cardiac valve disease, HFrEF (LVEF <45%), asthma.
* Previous stroke or significant neurological disease including cognitive dysfunction.
* Ongoing depression.
* Hypothyroidism
* Unable or unwilling to participate in training, e.g., due to injury, arthrosis or lung disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants >60 years.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
[15O]H2O PET assessment of the blood perfusion of the brain | 2 years
  We will use the scan to determine our primary outcome: Blood perfusion to the heart and brain.
  Radioactive water ([15O]H2O) will be used as a PET-tracer since it follows the blood and is the gold standard tracer for PET-based blood perfusion measurements.
  We measure the blood perfusion of the brain as the perfusion capacity, meaning the difference between blood perfusion to the organ at rest and the maximally possible perfusion. In the brain we use injection of diamox to stimualte maximal dilation of the cerebral arteries which corresponds to the maximally possible perfusion of the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas EHJ Primary Investigator, Medical Doctor, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Have not gotten the necessary clearence